CLINICAL TRIAL: NCT06879847
Title: A Single-arm, Prospective Clinical Study on the Efficacy of Total Body Irradiation Combined with Busulfan and Melphalan As Conditioning Regimen for Patients with Relapsed/Refractory Acute Myeloid Leukemia Undergoing Salvage HSCT
Brief Title: A Single-arm, Prospective Study of TBI + BUMEL As a Conditioning Regimen for Salvage HSCT in Patients with R/R AML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-WXJ-2024-475
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia
Keywords: Salvage Allogeneic Hematopoietic Stem Cell Transplantation; Relapsed or Refractory Acute Myeloid Leukemia; Conditioning Regimen; Total Body Irradiation; Melphalan
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 40 patients with relapsed/refractory acute myeloid leukemia who undergo HSCT (Experimental): patients undergo HSCT using TBI + BUMEL as a conditioning regimen
  Interventions: Procedure: Salvage Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Salvage Allogeneic Hematopoietic Stem Cell Transplantation — 1. TBI+BUMEL (IBM) Conditioning Regimen Day -7: Semustine (Me-CCNU) 250mg/m², orally, Day -7; Day -6: Total Body Irradiation (TBI) 4Gy, in two parts, Day -6; Day -5 to Day -4: Busulfan (Bu) 3.2mg/kg/day, administered in four divided doses, IV infusion; Day -3 to Day -2: Melphalan (Mel) 50mg/m²/day, IV infusion
  2. Donor Stem Cell Infusion (Hematopoietic Stem Cell Transplantation) Day 0: Intravenous infusion of donor hematopoietic stem cells (MNC ≥ 8×10⁸/kg, CD34+ cells ≥ 4×10⁶/kg).

SUMMARY:
Acute myeloid leukemia (AML) is one of the hematologic malignancies, for which patients typically undergo chemotherapy to achieve complete remission. However, approximately 30% of patients fail to respond to initial treatment, and many experience relapse after achieving remission. For patients with relapsed or refractory AML, allogeneic hematopoietic stem cell transplantation (HSCT) offers a potentially curative option. Sibling-matched HSCT has demonstrated a disease-free survival rate of 20-30%, while unrelated donor transplants yield an overall survival rate of approximately 22%. Haploidentical transplantation is a viable alternative for patients lacking a sibling donor. A 2019 study involving 1,693 patients with relapsed/refractory (R/R) AML revealed that haploidentical transplants yielded outcomes comparable to other transplant modalities, including HLA-matched and 9/10 matched unrelated donor transplants, thus supporting haploidentical transplantation as a viable therapeutic option.

The conditioning regimen is a critical component of the transplantation. In China, the modified BU/CY conditioning regimen, which combines busulfan (BU) and cyclophosphamide (CTX), is widely utilized for tumor cytoreduction and immunosuppression. Some centers also employ post-transplant cyclophosphamide (PTCy) to mitigate the risk of graft-versus-host disease (GVHD). Despite advances, relapse remains a significant challenge. Optimizing conditioning regimens to enhance tumor cell targeting and achieve deeper remission is crucial. Additionally, many patients are unfit due to prior chemotherapy, infections, and organ dysfunction, which may make them unable to tolerate high-intensity conditioning.

Recent studies suggest that melphalan (MEL)-based conditioning regimens may offer advantages over CTX-based protocols. While total body irradiation (TBI) has been traditionally used in conditioning for HSCT, it is associated with considerable organ toxicity.

A low-dose TBI regimen combined with BU+MEL represents a promising conditioning regimen for R/R AML. In preliminary studies, 7 patients treated with this regimen successfully achieved hematopoietic stem cell engraftment. Building on these results, a clinical study is planned to evaluate further the safety and efficacy of the TBI+BUMEL (IBM) conditioning regimen in relapsed/refractory AML, with a focus on improving engraftment rates, reducing relapse rates, minimizing GVHD incidence, and enhancing overall survival outcomes.

DETAILED DESCRIPTION:
The aim of this study is to observe the efficacy-related factors and adverse events of the TBI combined with BUMEL regimen as conditioning for allogeneic hematopoietic stem cell transplantation in patients with relapsed/refractory acute myeloid leukemia .

ELIGIBILITY:
Inclusion Criteria:

1. Age between 14 and 70 years (inclusive of the age limits);
2. Patients diagnosed with relapsed/refractory (R/R) AML, meeting the World Health Organization (WHO) 2016 AML diagnostic criteria, must meet one of the following definitions:

   Relapsed AML: Leukemic cells reappear in peripheral blood or bone marrow blasts >5% after achieving complete remission (CR, CRi) (excluding other causes such as bone marrow regeneration following consolidation chemotherapy), or extramedullary leukemic infiltration occurs.

   Refractory AML:Initial cases that do not respond to two courses of standard treatment. Relapse within 12 months after consolidation therapy. Relapse after 12 months with no response to conventional chemotherapy. Two or more relapses. Persistent extramedullary leukemia.
3. Heart, liver, and kidney function must meet the following criteria:

   Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 3× the upper limit of normal (ULN); Total bilirubin ≤ 3× ULN; Serum creatinine ≤ 2× ULN or creatinine clearance ≥ 40 mL/min; Left ventricular ejection fraction (LVEF), as measured by echocardiography or multi-gated acquisition (MUGA) scan, must be within the normal range (>50%).
4. Availability of a suitable allogeneic donor;
5. Life expectancy of ≥3 months;
6. Karnofsky Performance Status (KPS) ≥ 60%, Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
7. The patient understands the study protocol and voluntarily signs the informed consent form.

Exclusion Criteria:

1. Patients had serious adverse reactions to investigational drugs such as allergies;
2. Patients with a history of immunodeficiency, or other acquired or congenital diseases, immunodeficiency diseases, and a history of organ transplantation;
3. Patients with hypertension, ventricular arrhythmia requiring clinical intervention, acute coronary syndrome, congestive heart failure, stroke, or other grade III or higher cardiovascular events within 6 months;
4. Patients received Class II or higher surgery within 4 weeks prior to enrollment;
5. Patient has an active and difficult-to-control infection, including but not limited to active fungal, bacterial, or viral infections that require systemic treatment, such as active HIV, hepatitis B or C;
6. Patient has active central nervous system leukemia infiltration;
7. Pregnant or lactating patients;
8. Patient is currently participating in another clinical studies;
9. Other conditions where the investigator deems the patient unsuitable for inclusion.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidence of neutrophil engraftment and platelet engraftment | on day 28±7 following HSCT
  Neutrophil and platelet engraftment is defined as the first occurrence of 3 consecutive days with an absolute neutrophil count of at least 0.5×109/L and a platelet count of over 20×109/L for 7 consecutive days without transfusion support.
The time to reconstitution of hematopoiesis | on day 28±7 following HSCT
  recovery of hemopoietic function after treatment
The cumulative incidence of transplant-related mortality (TRM) | within 100 days following HSCT
  Transplant-related mortality was defined as mortality due to any cause other than disease progression within 100 days of transplantation.

SECONDARY OUTCOMES:
The cumulative incidence and grade of graft-versus-host disease (GVHD) | within 1 year following HSCT
  Graft-versus-host disease (GVHD) is a medical complication following the receipt of transplanted tissue from a genetically different person.
The cumulative incidence of relapse | within 1 year following HSCT
  We defined relapse as any clinical evidence of progression or recurrence of original diseases.
Overall survival rate | within 1 year following HSCT
  We estimated OS from the time of transplant until the date of death of any cause or last follow-up for patients still alive.
The cumulative incidence of adverse events | within 1 year following HSCT
  Following extraction of the tumor, a blood vessel burst causing increased blood loss during the procedure, an adverse event the surgeon did not expect.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, Prof., Study Chair — The First Affiliated Hospital of Soochow University; Xiaojin Wu, Prof., Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- Hematology Department, The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No